CLINICAL TRIAL: NCT01319838
Title: Prolonged Isotretinoin Therapy in Patients With High Risk Neuroblastoma
Brief Title: Aflac ST1001 Prolonged Isotretinoin
Acronym: Aflac ST1001
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: no patient enrollment
Sponsor: Emory University (Other)
Collaborators: Children's Healthcare of Atlanta (Other)
Responsible Party: Principal Investigator, Muna Qayed, Principal Investigator, Emory University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00047148; Aflac ST1001 (Other: Other)
Record Dates: First submitted 2011-03-18; First posted 2011-03-22 (Estimated); Last update posted 2013-12-10 (Estimated); Status verified 2013-12

CONDITIONS: Neuroblastoma
Keywords: neuroblastoma; isotretinoin
MeSH Terms: conditions — Neuroblastoma | interventions — Isotretinoin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- isotretinoin prolongation (Experimental): Prolonged treatment with isotretinoin, extending standard 6 month duration to 2 years
  Interventions: Drug: Isotretinoin

INTERVENTIONS:
Drug: Isotretinoin — >12 kg: 160 mg/m2/day, given PO, divided BID <=12 kg: 5.33 mg/kg/day, given PO, dividied BID doses given days 1-14 of 28 day cycle for 24 consecutive cycles

SUMMARY:
Neuroblastoma is a cancer of the nervous system and accounts for 15% of cancer related deaths in children. With the advancement of treatment therapies, the long term survival rate has progressed to approximately 50%. The therapy used for treatment, however, is very toxic and associated with serious long-term side effects. Treatment for neuroblastoma typically includes chemotherapy, surgery, stem cell transplantation, radiation therapy, and immunotherapy. At the end of this treatment, children with neuroblastoma commonly take the drug isotretinoin for 6 months. Isotretinoin maintains the response to previous treatments and helps turn the remaining cancer cells into normal nerve cells.

Most patients often respond to this treatment at first but are at a high-risk for the cancer coming back. The majority of the children who relapse after treatment or develop recurrent disease do so in the first two years following the completion of therapy and there are no current treatments to cure those who relapse. This study will explore whether or not extending the therapy with isotretinoin from 6 months to 24 months will help prevent the cancer from coming back without causing severe side effects.

DETAILED DESCRIPTION:
Neuroblastoma is the most common extracranial solid tumor of childhood and accounts for 15% of all pediatric cancer related deaths. The majority of patients present with high-risk disease that is widely metastatic and aggressive. Historically, less than 30% of these patients achieved long-term disease-free survival and the majority of relapses occurred within the first 24 months following treatment. Survival rates have modestly improved with the addition of high-dose chemotherapy and stem cell rescue, radiotherapy, surgery and biologic therapy, yet 50% of patients still succumb to their disease. Current treatment of neuroblastoma also carries significant acute toxicities and those patients that are cured suffer significant long-term treatment-related morbidities. Therefore, children with high-risk neuroblastoma are in need of novel therapeutic strategies that will improve cure rates without adding to acute and long-term toxicities.

Retinoids, derivatives of vitamin A, have been repeatedly shown to arrest cell growth of neuroblastoma cells in vitro by causing differentiation. Clinical trials in relapsed neuroblastoma patients with bulky tumors failed to show significant responses to retinoid therapy. Subsequently, however, a sentinel randomized clinical trial demonstrated that isotretinoin(13-cis-retinoic acid), when given to patients with minimal residual disease following consolidation chemotherapy, independently improved the overall survival of patients with high-risk neuroblastoma. The treatment regimen included isotretinoin for 2 weeks followed by a 2 week rest period for 6 treatment cycles. The treatment was very well tolerated with minimal side effects. The duration of treatment, 6 months, was arbitrarily chosen and currently many institutions implement prolonged retinoic acid treatment in patients with relapsed high-risk disease, yet no formal study has been done to statistically show improved survival with prolonged biotherapy.

To improve the progression-free survival in patients with high-risk neuroblastoma this trial will prolong therapy with isotretinoin to 24 months, the time window in which most relapses occur. The treatment is anticipated to be well tolerated with no increase in adverse side effects based on the benign side effect profile of patients who have received the typical 6 month treatment course. The trial will consist of a single arm of 20 high-risk neuroblastoma patients who will receive a total of 24 cycles of isotretinoin (2 weeks on treatment followed by 2 weeks of rest) compared to the historical and current COG study treatment of 6 cycles. Patients will be accrued over a 3-year period.

The toxicity and tolerability of a prolonged course of isotretinoin biologic therapy will be closely monitored with a focus on neuropsychologic and bone toxicities, and isotretinoin drug levels will be measured to determine if there is a correlation between levels and anti-tumor efficacy or toxicities. This will provide complementary data to support future national cooperative group trials.

ELIGIBILITY:
Inclusion Criteria:

* <=30 years of age
* histologic verification of neuroblastoma
* no active measurable disease on CT/MRI
* ultra high risk status by having mixed response, no response or stable disease following initial treatment or by having recurrent neuroblastoma
* Karnofsky >=50% for patients >16 years and Lansky >=50% for patients <=16 years
* patients must have completed high risk therapy
* organ function as defined in protocol

Exclusion Criteria:

* patients with active measurable disease
* patients who are pregnant or breast-feeding
* concomitant medications stopped as indicated in protocol
* patients with uncontrolled infection
* patients with history of depression or psychotic disorder requiring medication

Max Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2011-03; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Progression free survival | 5 years after treatment completed
  To determine the progression free survival in patients with high risk neuroblastoma who receive a prolonged course of biologic therapy with isotretinoin
Isotretinoin toxicity | 5 years after treatment completed
  To determine the toxicity and tolerability of a prolonged course of isotretinoin biologic therapy

SECONDARY OUTCOMES:
Bone growth effect | 5 years after treatment completed
  To observe any effects on bone growth and metabolism in patients receiving a prolonged course of isotretinoin biologic therapy
Isotretinoin pharmacokinetic profile | 1 year after treatment completed
  To determine changes in time of the pharmacokinetic profile of a prolonged course of isotretinoin biologic immunotherapy
Neurologic or psychologic sequelae | 1 year after treatment completed
  To observe the incidence of neurologic or psychologic sequelae resulting from a prolonged course of isotretinoin biologic therapy

CONTACTS AND LOCATIONS:
Overall Officials: Howard Katzenstein, MD, Principal Investigator — Children's Healthcare of Atlanta/Emory University
Locations (1):
- Children's Healthcare of Atlanta, Atlanta, Georgia, United States

REFERENCES:
- See also: clinical trials website — http://www.choa.org/Childrens-Hospital-Services/Cancer-and-Blood-Disorders/Research/Clinical-Trials/Find-a-Clinical-Trial